CLINICAL TRIAL: NCT03363984
Title: A Single-center, Open-label Study to Investigate the Effect of a Single Oral Dose and Repeated Oral Doses of ID-082 on the Pharmacokinetics of Midazolam and Its Metabolite 1-hydroxymidazolam in Healthy Male Subjects.
Brief Title: Pharmacokinetic Interaction Between Midazolam and ID-082 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID-082-102
Record Dates: First submitted 2017-11-21; First posted 2017-12-06 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midazolam & ID-082 (Experimental): Single oral administration of 2 mg midazolam on Day 1, Day 2, and Day 11. Administration of ID-082 from Day 2 through Day 11.
  Interventions: Drug: Midazolam; Drug: ID-082

INTERVENTIONS:
Drug: Midazolam — Single oral administration of 2 mg midazolam under fasted conditions/outside of meal times
Drug: ID-082 — Administration of ID-082 under fasted conditions/outside of meal times

SUMMARY:
A clinical study in healthy male subjects to investigate whether the administration of ID-082 can affect the fate in the body (amount and time of presence in the blood) of midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure;
* Healthy male subjects aged 18 to 45 years (inclusive) at screening;
* Male subject with a female partner of childbearing potential or a pregnant partner must agree to use a condom from screening, during the study, and for at least 3 months after last study treatment intake;
* Body mass index of 18.0 to 30.0 kg/m2 (inclusive) at screening;
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests.

Exclusion Criteria:

* Contraindication or known hypersensitivity to ID-082, midazolam or drugs of the same classes, or any of their excipients;
* Modified Swiss Narcolepsy Scale total score < 0 at Screening or history of narcolepsy or cataplexy;
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study treatment;
* Known hypersensitivity or allergy to natural rubber latex;
* Known hereditary problems of fructose intolerance, glucose-galactose malabsorption, or sucrose-isomaltase insufficiency;
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions;
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Cmax of midazolam | From baseline to EOS (i.e. for up to 16 days)
  Maximum plasma concentration
AUC0-24 of midazolam | From baseline to EOS (i.e. for up to 16 days)
  Area under the plasma concentration-time curvefrom time zero to 24 h

SECONDARY OUTCOMES:
Cmax of 1-hydroxymidazolam | From baseline to EOS (i.e. for up to 16 days)
  Maximum plasma concentration
AUC0-inf of midazolam and 1-hydroxymidazolam and AUC0-24 of 1-hydroxymidazolam | From baseline to EOS (i.e. for up to 16 days)
  Area under the plasma concentration-time curve from zero to infinity
tmax of midazolam and 1-hydroxymidazolam | From baseline to EOS (i.e. for up to 16 days)
  Time to reach maximum plasma concentration
t½ of midazolam and 1-hydroxymidazolam | From baseline to EOS (i.e. for up to 16 days)
  Terminal elimination half-life
Total body apparent plasma clearance (CL/F) of midazolam | From baseline to EOS (i.e. for up to 16 days)
Metabolic ratio (MR) of the AUC0-24 of 1-hydroxymidazolam to the AUC0-24 of midazolam | From baseline to EOS (i.e. for up to 16 days)

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Le Gac, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, Mid Galmorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: No